CLINICAL TRIAL: NCT04353817
Title: A Phase 3b, Randomized, Placebo-controlled Study Evaluating the Efficacy and Safety of Elexacaftor/Tezacaftor/Ivacaftor in Cystic Fibrosis Subjects 6 Through 11 Years of Age Who Are Heterozygous for the F508del Mutation and a Minimal Function Mutation (F/MF)
Brief Title: A Study Evaluating Efficacy and Safety of Elexacaftor/Tezacaftor/Ivacaftor in Subjects 6 Through 11 Years of Age With Cystic Fibrosis and F/MF Genotypes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX19-445-116; 2019-003554-86 (EudraCT Number)
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Results first posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo matched to ELX/TEZ/IVA and placebo matched to IVA in the treatment period for 24 weeks.
  Interventions: Other: Placebo (matched to ELX/TEZ/IVA); Other: Placebo (matched to IVA)
- ELX/TEZ/IVA (Experimental): Participants weighing less than (<) 30 kilograms (kg) at screening received ELX 100 mg qd/TEZ 50 mg qd/IVA 75 mg every 12 hours (q12h) and participants weighing greater than equals to (>=) 30 kg at screening received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 24 weeks.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed-dose combination tablet for oral administration qd in the morning.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
  Arms: ELX/TEZ/IVA
Drug: IVA — Tablet for oral administration qd in the evening.
  Other Names: VX-770; ivacaftor
  Arms: ELX/TEZ/IVA
Other: Placebo (matched to ELX/TEZ/IVA) — Placebo matched to ELX/TEZ/IVA for oral administration once daily (qd) in the morning.
  Arms: Placebo
Other: Placebo (matched to IVA) — Placebo matched to IVA for oral administration qd in the evening.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of elexacaftor (ELX) / tezacaftor (TEZ) / ivacaftor (IVA) triple combination (TC) in subjects 6 through 11 years of age with cystic fibrosis (CF) who are heterozygous for F508del and a minimal function (MF) mutation (F/MF genotypes).

ELIGIBILITY:
Key Inclusion Criteria:

* Heterozygous for the F508del mutation (F/MF)
* Forced expiratory volume in 1 second (FEV1) value greater than equal to(≥) 70%

Key Exclusion Criteria:

* Clinically significant cirrhosis with or without portal hypertension
* Lung infection with organisms associated with a more rapid decline in pulmonary status
* Solid organ or hematological transplantation

Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- Australia (3):
  - Telethon Kids Institute, Nedlands
  - Queensland Children's Hospital, South Brisbane
  - The Children's Hospital at Westmead, Westmead
- Canada (3):
  - McGill University Health Centre, Glen Site, Montreal Children's Hospital, Montreal
  - The Hospital for Sick Children, Toronto
  - British Columbia Children's Hospital, Vancouver
- Juliane Marie Center, Rigshospitalet, Copenhagen, Denmark
- France (5):
  - Groupe Hospitaler Pellegrin, CHU De Bordeaux, Bordeaux
  - CHU Lyon - Hopital Femme Mere-Enfant, Bron
  - Hopital Necker, Enfants Malades, Paris
  - Hopital Robert Debre, Paris
  - Centre de Perharidy, Roscoff
- Germany (7):
  - Charite Paediatric Pulmonology Department, Berlin
  - Universitaetsklinkum Koeln, CF-Studienzentrum, Cologne
  - Universitätsklinikum Essen, Essen
  - Johann Wolfgang Goethe University, Frankfurt
  - Justus-Liebig-Universität Gießen Zentrum fur Kinderheilkunde und Jugendmedizin, Giessen
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Heidelberg, Zenter fuer Kinder-und Jugendmedizin, Heidelberg
- Israel (2):
  - Hadassah University Hospital Mount Scopus, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - Erasmus Medical Center / Sophia Children's Hospital, Rotterdam
- Spain (2):
  - Hospital Universitari Vall d Hebron, Barcelona
  - Hospital Virgen de la Arrixaca, Murcia
- Switzerland (2):
  - Inselspital - Universitaetsspital Bern, Bern
  - Kinderspital Zuerich, Zurich
- United Kingdom (7):
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol Royal Hospital, Bristol
  - Children's Hospital of Wales, Cardiff
  - Royal Hospital for Sick Children, Edinburgh
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Great Ormond Street Hospital for Sick Children, London
  - Royal Brompton & Harefield NHS Foundation Trust, Royal Brompton Hospital, London
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted in cystic fibrosis (CF) participants aged 6 through 11 years of age.
Groups:
- ELX/TEZ/IVA: Participants weighing less than (<) 30 kilograms (kg) at screening received ELX 100 mg once daily (qd)/TEZ 50 mg qd/IVA 75 mg every 12 hours (q12h) and participants weighing greater than equals to (>=) 30 kg at screening received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 24 weeks.
Period: Overall Study
Arm/Group | Placebo | ELX/TEZ/IVA
Started | 61 | 60
Completed | 61 | 59
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- ELX/TEZ/IVA: Participants weighing <30 kg at screening received ELX 100 mg qd/TEZ 50 mg qd/IVA 75 mg q12h and participants weighing >=30 kg at screening received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | ELX/TEZ/IVA | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.2 (1.7) | 9.1 (1.8) | 9.2 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 26 | 25 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 42 | 48 | 90
  Unknown or Not Reported | 19 | 11 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 42 | 45 | 87
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 19 | 11 | 30
Lung Clearance Index2.5 (LCI2.5) [Mean (Standard Deviation); unit: index] — The LCI2.5 index is the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/40th of its starting values and is calculated by dividing the sum of exhaled tidal breaths (cumulative exhaled volume (CEV)) by simultaneously measured functional residual capacity (FRC). An LCI of 7.5 and below is normal; values greater than 7.5 are abnormal. LCI is able to detect abnormalities in lung function earlier than more traditional modalities such as spirometry.
  index | 9.75 (1.95) | 10.26 (2.22) | 10.01 (2.09)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Lung Clearance Index 2.5 (LCI2.5)
Description: The LCI2.5 index is the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/40th of its starting values and is calculated by dividing the sum of exhaled tidal breaths (cumulative exhaled volume (CEV)) by simultaneously measured functional residual capacity (FRC). An LCI of 7.5 and below is normal; values greater than 7.5 are abnormal. LCI is able to detect abnormalities in lung function earlier than more traditional modalities such as spirometry.
Time Frame: From Baseline Through Week 24
Population: Full analysis set (FAS) included all randomized participants who carry the intended CFTR allele mutation and receive at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: index
Arm/Group | Placebo | ELX/TEZ/IVA
Number analyzed (Participants) | 61 | 60
index | -0.02 (0.16) | -2.29 (0.16)
Statistical Analysis 1: Comparison: Placebo vs ELX/TEZ/IVA; Test type: Superiority; p < 0.0001, Mixed-effects Model for Repeated Measure; Least Squares (LS) Mean Difference = -2.26, 95% CI 2-sided [-2.71 to -1.81]

2. Secondary Outcome: Absolute Change in Sweat Chloride (SwCl)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline Through Week 24
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | Placebo | ELX/TEZ/IVA
Number analyzed (Participants) | 61 | 60
millimole per liter (mmol/L) | -0.9 (1.5) | -52.1 (1.5)
Statistical Analysis 1: Comparison: Placebo vs ELX/TEZ/IVA; Test type: Superiority; p < 0.0001, Mixed-effects Model for Repeated Measure — This is the nominal p-value without multiplicity controlled; LS Mean Difference = -51.2, 95% CI 2-sided [-55.3 to -47.1]

3. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 28
Population: Safety set included all participants who received at least 1 dose of study drug in the treatment period.
Measure: Number; unit: participants
Arm/Group | Placebo | ELX/TEZ/IVA
Number analyzed (Participants) | 61 | 60
participants
  Participants With TEAEs | 57 | 48
  Participants With SAEs | 9 | 4

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 28
Arm/Group | Placebo | ELX/TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/60
Serious Adverse Events (participants affected / at risk) | 9/61 | 4/60
Other Adverse Events (participants affected / at risk) | 53/61 | 46/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=61) | ELX/TEZ/IVA (N=60)
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 3 | 0
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 1
Bacterial test positive (Investigations) | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=61) | ELX/TEZ/IVA (N=60)
Abdominal pain (Gastrointestinal disorders) | 17 | 5
Abdominal pain upper (Gastrointestinal disorders) | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Nausea (Gastrointestinal disorders) | 5 | 1
Steatorrhoea (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 4 | 3
Fatigue (General disorders) | 5 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 14 | 1
Nasopharyngitis (Infections and infestations) | 9 | 7
Rhinitis (Infections and infestations) | 5 | 3
Upper respiratory tract infection (Infections and infestations) | 5 | 3
Alanine aminotransferase increased (Investigations) | 3 | 5
Aspartate aminotransferase increased (Investigations) | 1 | 3
Bacterial test positive (Investigations) | 4 | 0
Forced expiratory volume decreased (Investigations) | 4 | 0
Staphylococcus test positive (Investigations) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Headache (Nervous system disorders) | 12 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 14
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT04353817/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT04353817/SAP_001.pdf